CLINICAL TRIAL: NCT00977002
Title: Prevention of Reintubation by Using Noninvasive Positive Pressure Ventilation: Randomized Controlled Trial
Brief Title: Prevention of Reintubation by Using Noninvasive Positive Pressure Ventilation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: Rafaelle Fernandes Batistella, UNESP- Botucatu Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: upeclin/HC/FMB-Unesp-23
Record Dates: First submitted 2009-09-14; First posted 2009-09-15 (Estimated); Last update posted 2011-02-02 (Estimated); Status verified 2011-02

CONDITIONS: Extubation Failure; Acute Respiratory Failure Post Extubation
Keywords: noninvasive ventilation; extubation; Respiratory failure; reintubation
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Noninvasive Ventilation; Oxygen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- PPNIV (Experimental): Patient randomized to this group will be ventilated with Positive Pressure Noninvasive Ventilation post extubation
  Interventions: Other: Positive Pressure Noninvasive ventilation
- O2I (Active Comparator): Patient randomized to this group will be submitted to traditional oxygen therapy post extubation
  Interventions: Other: Inhalatory O2

INTERVENTIONS:
Other: Positive Pressure Noninvasive ventilation — Patients randomized to this group are submitted to positive pressure noninvasive ventilation for 12 hours or more. Children younger than one year use nasal prong and older than one year use nasal or facial mask. A blood gas is collected in the moment of intubation and one hour after.
  Other Names: Noninvasive ventilation
  Arms: PPNIV
Other: Inhalatory O2 — Patients randomized to this group are submitted to inhalatory O2 using mask or nasal catheter. A blood gas is collected in the moment of intubation and one hour after.
  Other Names: Oxygen therapy
  Arms: O2I

SUMMARY:
Child extubation failure range from 4.1% to 19%. Studies in adults and children showed that extubation failure increases mortality mainly in those who need reintubation as this is a invasive procedure associated with many complications. Therefore, patients are reintubated when they worsen, which can contribute to organ dysfunction and increased mortality.

Positive Pressure Noninvasive ventilation (PPNIV) has been proposed as a way to treat acute respiratory distress, avoiding complications of intubation and invasive ventilation. Most of the studies in adults are not conclusive on the benefits of PPNIV as a way to treat post-extubation acute respiratory distress. However, studies that evaluated the early use of PPNIV in post-extubation period as a way to prevent respiratory failure tend to show some advantages as decrease of reintubation, decrease number of respiratory distress, decrease of hospital infection frequency and lower mortality rate in the intensive care unit (ICU) for those who use PPNIV.

In a prospective study on the use of PPNIV in 114 children, Essouri at al avoided invasive ventilation in 77%, being the group in patients with post-extubation respiratory distress.

As far as the investigators know there is not any randomized, controlled study in children examining the PPNIV as a way to prevent post-extubation respiratory distress. The investigators' hypothesis is that PPNIV decreases the extubation failure rate and, as a consequence, the Pediatric Intensive Care Unit (PICU) and hospital length of stay, and mortality rate.

The objective is to compare PPNIV and inhalatory O2 (catheter or facial mask) in children after extubation, evaluating the need of reintubation, hospital and PICU mortality rate and length of stay in PICU and hospital.

DETAILED DESCRIPTION:
Prospective, randomized and controlled study at the PICU - University Hospital, Botucatu Medical School-UNESP. Patients elegibled are exposed to extubation test. If passed they are randomized in two groups: 1) post-extubation PPNIV (PPNIV, n=50), and 2) Inhalatory oxygen therapy by nasal catheter or facial mask (O2I, n=50). Patients are observed for 48 hours, being considered extubation failure if they need reintubation. Arterial blood gas is obtained at the day or programed extubation and one hour after extubation.

Nasal prongs and facial or nasal masks are used in accordance with child age. All patients from this group are kept in PPNIV for a 12 hours at least. Feeding, if released, is done by gastric probe.

In O2IG, patients use facial mask or nasal catheter after extubation. Both groups are submitted to physiotherapy and nurse care as the PICU routine Follow up: Variables: age, gender, disease and comorbidities, intubation cause , time intubated and invasive ventilation use, PRISM score at the moment of admission, risk factors to respiratory distress post extubation, Comfort scale just before extubation, use of sedatives (time and mean dose)during invasive ventilation. At randomization and one hour later: vital signs, arterial blood gas. Patients are followed for 48 hour to evaluate reintubation and then for other complications, death and length of stay in PICU and hospital.

ELIGIBILITY:
Inclusion Criteria:

Patients aged between 28 days and 15 years and who were intubated and remained under invasive mechanical ventilation for 48 hours, passed in the extubation test for, and who presented at least one of the following risk factors for respiratory distress post extubation:

1. Invasive ventilation for at least 15 days
2. Use of inotropics for more than 48 hours
3. Endovenous continuous administration of sedative/analgesic drugs
4. 1-3 months old
5. Mean Airway Pressure(Paw)> 8,5; Inspired fraction of O2(FiO2)> 0,4; Oxygenation index(IO)> 4,5 immediately before extubation
6. Cardiac or pulmonary chronic diseases
7. Cardiac output
8. Hipercapny: Arterial pressure of CO2 (PaCO2)> 45 mmHg

Exclusion Criteria:

1. Tracheostomized
2. Accidental extubation
3. Respiratory failure just after extubation, needing immediate reintubation
4. Neuromuscular diseases
5. Death
6. PPNIV exclusion: coma or disability to protect airway, not tolerated, hemodynamic instability, shock, cardiac disritmy, facial or intracranial traumatic injury or surgery that preclude use of mask, abdominal distension, nausea or vomiting, gastric or esophagic recent surgery, gastrointestinal hemorrhagy in activity, not drained pneumothorax.
7. Reintubated patients during its stay in PICU, that have already participated in this study

Ages: 28 Days to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Prevention of reintubation | 48 hours

SECONDARY OUTCOMES:
decrease of PICU and hospital mortality | 28 days
decrease of hospital and PICU length of stay | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Rafaelle F Batistella, Principal Investigator — FMB - UNESP; José R Fioretto, Study Director — FMB-UNESP; Mário F Carpi, Study Chair — FMB-UNESP
Locations (1):
- Botucatu Medical School-UNESP, Botucatu, São Paulo, Brazil